CLINICAL TRIAL: NCT02175004
Title: An Open-Label Extension Study to Assess the Long-Term Safety and Efficacy of ISIS 420915 in Patients With Familial Amyloid Polyneuropathy (FAP)
Brief Title: Extension Study Assessing Long Term Safety and Efficacy of IONIS-TTR Rx in Familial Amyloid Polyneuropathy (FAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 420915-CS3; 2013-004561-13 (EudraCT Number)
Expanded Access: NCT03400098 (Approved for marketing)
Record Dates: First submitted 2014-06-12; First posted 2014-06-26 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: FAP; Familial Amyloid Polyneuropathy; TTR; Transthyretin; Amyloidosis
Keywords: FAP; Familial Amyloid Polyneuropathy; TTR; Transthyretin; Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis | interventions — Inotersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Previous Placebo-Inotersen 300 mg (Experimental): Participants received subcutaneous (SC) doses of 300 milligrams (mg) inotersen once weekly for up to 260 weeks. Participants who received inotersen-matching placebo in the previous study- ISIS 420915-CS2 (NCT01737398) were included in this group.
  Interventions: Drug: Inotersen
- Previous Inotersen-Inotersen 300 mg (Experimental): Participants received SC doses of 300 mg inotersen once weekly for up to 260 weeks. Participants who received inotersen in the previous study- ISIS 420915-CS2 were included in this group.
  Interventions: Drug: Inotersen

INTERVENTIONS:
Drug: Inotersen — Inotersen SC
  Other Names: TEGSEDI; IONIS-TTR Rx; ISIS 420915

SUMMARY:
This study evaluates the safety and tolerability of extended dosing with IONIS-TTR Rx in patients with Familial Amyloid Polyneuropathy.

DETAILED DESCRIPTION:
Familial Amyloid Polyneuropathy (FAP) is a rare, hereditary disease caused by mutations in the transthyretin (TTR) protein. TTR is made by the liver and secreted into the blood. TTR mutations cause it to misfold and deposit in multiple organs causing FAP.

IONIS-TTR Rx is an antisense drug that is designed to decrease the amount of mutant and normal TTR made by the liver. It is predicted that decreasing the amount of TTR protein will result in a decrease in the formation of TTR deposits, and thus slow or stop disease progression.

This study evaluates the safety and tolerability of extended dosing with IONIS-TTR Rx in patients with Familial Amyloid Polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory completion of dosing & efficacy assessments in ISIS 420915-CS2

Exclusion Criteria:

* Any new condition or worsening of existing condition that could make the patient unsuitable for participation, or interfere with the patient participating in and/or completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (9):
  - University of California, Irvine, Orange, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University Bayview Medical Center, Baltimore, Maryland
  - Boston University School of Medicine - Amyloid Treatment & Research Program, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center - The Neurological Institute, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
- FLENI, Buenos Aires, Argentina
- Brazil (2):
  - Federal University of Rio de Janeiro - University Hospital, Rio de Janeiro
  - AACD, São Paulo
- France (2):
  - CHU Henri Mondor - Department of Neurology, Créteil
  - CHU Bicetre Aphp French Referral Center for FAP/Cornamyl Network, Le Kremlin-Bicêtre
- UKM; Universitätsklinikum Münster, Klinik für Transplantationsmedizin, Münster, Germany
- Italy (2):
  - Universita Degli Studi Di Messina - Azienda Ospedaliera Universitaria Policlinico "Gaetano Martino", Messina, Sicily
  - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche - Fondazione IRCCS Policlinico San Matteo, Pavia
- Portugal (2):
  - CHLN - Hospital de Santa Maria, Lisbon
  - CHP-HGSA, Unidade Clinica de Paramiloidose, Porto
- Spain (2):
  - Hospital Universitari Vall D' Hebron, Barcelona
  - Hospital Clinic, Barcelona
- University College London - National Amyloidosis Centre, London, United Kingdom

REFERENCES:
- [Derived] Brannagan TH, Coelho T, Wang AK, Polydefkis MJ, Dyck PJ, Berk JL, Drachman B, Gorevic P, Whelan C, Conceicao I, Plante-Bordeneuve V, Merlini G, Obici L, Plana JMC, Gamez J, Kristen AV, Mazzeo A, Gentile L, Narayana A, Olugemo K, Aquino P, Benson MD, Gertz M; NEURO-T. T. R. Open-Label Extension Investigators. Long-term efficacy and safety of inotersen for hereditary transthyretin amyloidosis: NEURO-TTR open-label extension 3-year update. J Neurol. 2022 Dec;269(12):6416-6427. doi: 10.1007/s00415-022-11276-8. Epub 2022 Jul 31. PMID 35908242
- [Derived] Karam C, Brown D, Yang M, Done N, Zhu JJ, Greatsinger A, Bozas A, Vera-Llonch M, Signorovitch J. Long-term treatment effects of inotersen on health-related quality of life in patients with hATTR amyloidosis with polyneuropathy: Analysis of the open-label extension of the NEURO-TTR trial. Muscle Nerve. 2022 Oct;66(4):438-446. doi: 10.1002/mus.27675. Epub 2022 Aug 4. PMID 35799473
- [Derived] Yarlas A, Lovley A, McCausland K, Brown D, Vera-Llonch M, Conceicao I, Karam C, Khella S, Obici L, Waddington-Cruz M. Early Data on Long-term Impact of Inotersen on Quality-of-Life in Patients with Hereditary Transthyretin Amyloidosis Polyneuropathy: Open-Label Extension of NEURO-TTR. Neurol Ther. 2021 Dec;10(2):865-886. doi: 10.1007/s40120-021-00268-x. Epub 2021 Aug 5. PMID 34355354
- [Derived] Brannagan TH, Wang AK, Coelho T, Waddington Cruz M, Polydefkis MJ, Dyck PJ, Plante-Bordeneuve V, Berk JL, Barroso F, Merlini G, Conceicao I, Hughes SG, Kwoh J, Jung SW, Guthrie S, Pollock M, Benson MD, Gertz M; NEURO-TTR open-label extension investigators. Early data on long-term efficacy and safety of inotersen in patients with hereditary transthyretin amyloidosis: a 2-year update from the open-label extension of the NEURO-TTR trial. Eur J Neurol. 2020 Aug;27(8):1374-1381. doi: 10.1111/ene.14285. Epub 2020 May 29. PMID 32343462

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 135 participants, out of which 50 participants had received placebo, and 85 participants had received inotersen in the previous study ISIS 420915-CS2 (NCT01737398 - CS2 Study). Participants were enrolled into this study to receive inotersen. This study consisted of a 260-week Treatment Period, and a 3-month Post-treatment Evaluation Period. The data is reported as per the previous treatment received in CS2 study.
Period: Overall Study
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Started | 50 | 85
Completed | 9 | 9
Not Completed | 41 | 76
Not completed — Adverse Event or Serious Adverse Event (SAE) | 5 | 14
Not completed — Investigator Judgment | 1 | 4
Not completed — Voluntary Withdrawal | 6 | 19
Not completed — Liver Transplant | 1 | 0
Not completed — Disease Progression | 1 | 0
Not completed — Participants Started Treatment With Commercially Available/Post-study Inotersen | 27 | 39

BASELINE CHARACTERISTICS:
Population: Safety Set (SS) included all enrolled participants who received at least 1 injection of inotersen in Open-label Extension Study (ISIS 420915-CS3) (CS3).
Groups:
- Previous Placebo-Inotersen 300 mg: Participants received SC doses of 300 mg inotersen once weekly for up to 260 weeks. Participants who received inotersen-matching placebo in the previous study- ISIS 420915-CS2 were included in this group.
- Total: Total of all reporting groups
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg | Total
Number analyzed (Participants) | 50 | 85 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (14.62) | 60.3 (11.86) | 60.4 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 26 | 41
  Male | 35 | 59 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 44 | 73 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 0 | 3
  Race: Black | 0 | 1 | 1
  Race: White | 44 | 81 | 125
  Race: White & Grayish-Brown | 1 | 0 | 1
  Race: Other | 2 | 3 | 5
Percentage of Participants Abnormal Electroretinogram Results at Baseline [Number; unit: percentage of participants] — Population: Number analyzed is the number of participants with data available for analysis.
  percentage of participants
    number analyzed (Participants) | 39 | 76 | 115
    (all) | 51.3 | 18.4 | 29.6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Related to Study Drug
Description: An adverse event (AE) is any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. An SAE is any untoward medical occurrence that at any dose that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect, or is an important medical event. TEAEs considered related to the study drug as assessed by the Investigator are reported.
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
percentage of participants
  TEAEs | 100 | 96.5
  Serious TEAEs | 36.0 | 54.1
  TEAEs Related to Study Drug | 82.0 | 69.4

2. Primary Outcome: Percentage of Participants With Change From Baseline in Vital Signs
Description: Vital signs included blood pressure, heart rate, respiratory rate, and temperature. Only categories with at least one participant with event are reported.
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
percentage of participants
  Systolic Blood Pressure: <90 millimeters of mercury (mmHg) | 12.0 | 18.8
  Systolic Blood Pressure: >140 mmHg | 32.0 | 41.2
  Systolic Blood Pressure: >160 mmHg | 8.0 | 20.0
  Diastolic Blood Pressure: <50 mmHg | 6.0 | 9.4
  Diastolic Blood Pressure: >90 mmHg | 30.0 | 28.2
  Diastolic Blood Pressure: >100 mmHg | 10.0 | 7.1
  Heart Rate: <60 beats per minute (bpm) | 30.0 | 38.8
  Heart Rate: >100 bpm | 16.0 | 9.4
  Temperature (°C): <36.0°C | 46.0 | 55.3
  Respiratory Rate (breaths/minute): >20 breaths/minute | 24.0 | 21.2

3. Primary Outcome: Percentage of Participants With Change From Baseline in Weight
Description: As prespecified in the protocol, percentage of participants with change from baseline in weight is reported in 2 categories, decrease of ≥7% from Baseline and increase of ≥7% from Baseline.
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3. Overall number analyzed are the number of participants available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
percentage of participants
  Weight (kg): Decrease of ≥7% From Baseline | 30.0 | 47.1
  Weight (kg): Increase of ≥7% From Baseline | 24.0 | 11.8

4. Primary Outcome: Percentage of Participants With Clinically Significant Change From Baseline in Laboratory Test Values
Description: Clinical laboratory tests included the analysis of chemistry, haematology, and urinalysis. Any value outside the normal range will be flagged for the attention of the investigator who will assess whether or not a flagged value is of clinical significance. Only those categories with at least one participant with event are reported. Normal range of creatinine clearance is 110 to 150 mL/min in males and 100 to 130 mL/min in females. Normal urine protein to creatinine (P/C) ratio= <0.2. Normal range for Alanine Aminotransferase (ALT) is 4 to 36 units per liter (U/L). Platelets normal range=140×10^9/L to 400×10^9/L.
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3. Number analyzed is the number of participants with data available for analysis for the given category.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
percentage of participants
  Confirmed Creatinine Clearance by CKD-EPI <30 ml/min/1.73m^2 | 4.0 | 4.7
  Confirmed Urine P/C Ratio >5 × Upper Limit of Normal (ULN) | 8.0 | 10.6
  Confirmed Alanine Aminotransferase (ALT) ≥3 x ULN | 4.0 | 4.7
  Confirmed Value of Platelets <75 × 10^9/L | 12.0 | 12.9

5. Primary Outcome: Percentage of Participants With Change From Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF) as Determined by Electrocardiogram (ECG)
Description: Normal QTcF at Baseline is defined as ≤450 milliseconds (ms) for males or ≤470 ms for females. Percentage of participants with QT interval outside of normal range are reported.
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
percentage of participants
  QTcF >450 ms | 44.0 | 43.5
  QTcF >480 ms | 20.0 | 23.5
  QTcF >500 ms | 12.0 | 16.5

6. Primary Outcome: Percentage of Participants Using Concomitant Medication for Nervous and Cardiovascular System Disorders
Description: A concomitant therapy was any non-protocol-specified drug or substance (including over-the counter medications, herbal medications, and vitamin supplements) administered between signing of informed consent and the final post-treatment visit for treating nervous and cardiovascular system disorders.
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
percentage of participants
  Nervous System Disorders | 88.0 | 81.2
  Cardiovascular System Disorders | 68.0 | 75.3

7. Primary Outcome: Percentage of Participants With Change From Baseline in Ophthalmic Examination as Assessed by Visual Acuity Changes
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
percentage of participants | 0.0 | 2.4

8. Primary Outcome: Percentage of Participants With Change From Baseline in Light Detection Ability Measured by Electroretinography
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: SS included all enrolled participants who received at least 1 injection of inotersen in CS3. Overall number analyzed are the number of participants available for analyses. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 39 | 76
percentage of participants
  Participants With Change From Baseline at Week 78: number analyzed (Participants) | 28 | 63
  Participants With Change From Baseline at Week 78 | 25.0 | 12.7
  Participants With Change From Baseline at Week 156: number analyzed (Participants) | 16 | 33
  Participants With Change From Baseline at Week 156 | 31.3 | 9.1

9. Secondary Outcome: Change From Baseline in the Modified Neuropathy Impairment Score (mNIS)+7 Composite Score at Weeks 78 and 156
Description: The mNIS+7 composite score is a measure of neurologic impairment that evaluates muscle weakness, sensation, reflexes, nerve conduction, and autonomic function. The mNIS+7 Composite Score has a range of -22.32 to 346.32 and a higher mNIS+7 composite score indicates worsening disease. A positive change from Baseline indicates worsening of polyneuropathy impairments. Mixed Effects Model with Repeated Measures (MMRM) was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: Full Analysis Set (FAS) included all enrolled participants who received at least 1 injection of inotersen in this study (CS3) and who had at least 1 post-baseline efficacy assessment for the mNIS+7 score or Norfolk quality of life-diabetic neuropathy (QoL-DN) questionnaire total score collected after CS3 Study Day 1. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
score on a scale
  Change From Baseline at Week 78: number analyzed (Participants) | 31 | 66
  Change From Baseline at Week 78 | 33.11 (28.915) | 10.11 (18.204)
  Change From Baseline at Week 156: number analyzed (Participants) | 21 | 35
  Change From Baseline at Week 156 | 37.34 (29.030) | 17.21 (27.307)
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS+7 Composite Score at Week 78; Test type: Superiority; p < 0.001, MMRM — P-value= MMRM with fixed categorical effects for treatment, time, treatment-by-time interaction, each of 3 randomization stratification factors, fixed covariates for parent study baseline value, baseline-by-time interaction; Least Squares Mean Difference = -17.84, 95% CI 2-sided [-26.12 to -9.56]
Statistical Analysis 2: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS+7 Composite Score at Week 156; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -20.11, 95% CI 2-sided [-31.27 to -8.95]

10. Secondary Outcome: Change From Baseline in the mNIS +7 Component: Heart Rate to Deep Breathing Score at Weeks 78 and 156
Description: Heart rate to deep breathing is a quantitative autonomic test using the CASE IV instrument that measures a participant's change in heart rate after deep breathing. The score of this component ranges from 0 to 3.72 points. Higher scores indicate impairment. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: FAS included all enrolled participants who received at least 1 injection of inotersen in this study (CS3) and who had at least 1 post-baseline efficacy assessment for the mNIS+7 score or Norfolk QoL-DN questionnaire total score collected after CS3 Study Day 1. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
score on a scale
  Change From Baseline at Week 78: number analyzed (Participants) | 35 | 72
  Change From Baseline at Week 78 | 0.23 (0.977) | 0.11 (0.761)
  Change From Baseline at Week 156: number analyzed (Participants) | 22 | 39
  Change From Baseline at Week 156 | 0.44 (1.099) | 0.30 (0.504)
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Heart Rate to Deep Breathing Score at Week 78; Test type: Superiority; p = 0.638, MMRM — P-value=MMRM with fixed categorical effects for treatment, time, treatment-by-time interaction, each of 3 randomization stratification factors, fixed covariates for parent study baseline value, baseline-by-time interaction; Least Squares Mean Difference = -0.06, 95% CI 2-sided [-0.32 to 0.20]
Statistical Analysis 2: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Heart Rate to Deep Breathing Score at Week 156; Test type: Superiority; p = 0.965, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -0.01, 95% CI 2-sided [-0.30 to 0.29]

11. Secondary Outcome: Change From Baseline in the mNIS +7 Component: Nerve Conduction Score at Weeks 78 and 156
Description: The nerve conduction tests are quantitative tests that measure the conduction attributes of preselected nerves. The score range of this component is 0 to 18.6 points. Higher scores indicate impairment. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
score on a scale
  Change From Baseline at Week 78: number analyzed (Participants) | 32 | 68
  Change From Baseline at Week 78 | 1.86 (2.313) | 0.57 (1.361)
  Change From Baseline at Week 156: number analyzed (Participants) | 21 | 36
  Change From Baseline at Week 156 | 2.05 (2.351) | 0.77 (1.724)
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Nerve Conduction Score at Week 78; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -1.09, 95% CI 2-sided [-1.68 to -0.50]
Statistical Analysis 2: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Nerve Conduction Score at Week 156; Test type: Superiority; p = 0.067, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -0.66, 95% CI 2-sided [-1.38 to 0.05]

12. Secondary Outcome: Change From Baseline in the mNIS +7 Component: Heat-Pain Sensory Score at Weeks 78 and 156
Description: The Heat-Pain Sensory test uses the CASE IV instrument to perform standardized psychophysical measurement to determine pain sensory thresholds in response to heat. The maximum score of this component is 0 to 40 points. Higher scores indicate impairment. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
score on a scale
  Change From Baseline at Week 78: number analyzed (Participants) | 32 | 66
  Change From Baseline at Week 78 | 2.60 (8.440) | 2.45 (7.557)
  Change From Baseline at Week 156: number analyzed (Participants) | 21 | 35
  Change From Baseline at Week 156 | 2.90 (9.224) | 3.40 (8.774)
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Heat-Pain Sensory Score at Week 78; Test type: Superiority; p = 0.821, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = 0.34, 95% CI 2-sided [-2.67 to 3.36]
Statistical Analysis 2: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Heat-Pain Sensory Score at Week 156; Test type: Superiority; p = 0.293, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -2.16, 95% CI 2-sided [-6.21 to 1.90]

13. Secondary Outcome: Change From Baseline in the mNIS +7 Component: Touch-Pressure Sensory Score at Weeks 78 and 156
Description: The Touch-Pressure Sensory test uses the CASE IV instrument to perform standardized psychophysical measurement to determine pressure sensory thresholds in response to touch. The score range of this component is 0 to 40 points. Higher scores indicate impairment. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
score on a scale
  Change From Baseline at Week 78: number analyzed (Participants) | 32 | 66
  Change From Baseline at Week 78 | 1.00 (6.886) | -3.05 (8.878)
  Change From Baseline at Week 156: number analyzed (Participants) | 21 | 35
  Change From Baseline at Week 156 | 1.95 (6.866) | -2.34 (8.306)
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Touch-Pressure Sensory Score at Week 78; Test type: Superiority; p = 0.047, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -2.78, 95% CI 2-sided [-5.53 to -0.03]
Statistical Analysis 2: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the mNIS +7 Component: Touch-Pressure Sensory Score at Week 156; Test type: Superiority; p = 0.041, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -3.07, 95% CI 2-sided [-6.00 to -0.13]

14. Secondary Outcome: Change From Baseline in the Neuropathy Impairment (NIS) Composite Score at Week 52 of Years 4 and 5
Description: The NIS score is a measure of neurologic impairment. The NIS Score has a range of 0 to 244 and a higher NIS score indicates lower function. A positive change from Baseline indicates worsening. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Week 52 of Years 4 and 5
Population: FAS included all enrolled participants who received at least 1 injection of inotersen in this study (CS3) and who had at least 1 post-baseline efficacy assessment for the mNIS+7 score or Norfolk QoL-DN questionnaire total score collected after CS3 Study Day 1. Overall number analyzed are the number of participants available for analyses.Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 9 | 14
score on a scale
  Change From Baseline at Week 52 of Year 4 | 35.78 (21.071) | 18.32 (20.970)
  Change From Baseline at Week 52 of Year 5: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5 |  | 17.75 (NA) — Standard deviation (SD) was not estimable for 1 participant.
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the NIS Composite Score at Week 52 of Year 4; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -17.48, 95% CI 2-sided [-26.92 to -8.03]

15. Secondary Outcome: Change From Baseline in the NIS Component: Cranial Nerves Score at Week 52 of Years 4 and 5
Description: Cranial Nerve assessment involves testing 3rd and 6th nerves and facial, palate, and tongue weakness. The score range for this component is 0 to 40 points. Higher scores indicate worsening. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Week 52 of Years 4 and 5
Population: FAS included all enrolled participants who received at least 1 injection of inotersen in this study (CS3) and who had at least 1 post-baseline efficacy assessment for the mNIS+7 score or Norfolk QoL-DN questionnaire total score collected after CS3 Study Day 1. Overall number analyzed are the number of participants available for analyses. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 9 | 14
score on a scale
  Change From Baseline at Week 52 of Year 4 | 0.0 (0.0) | 0.0 (0.0)
  Change From Baseline at Week 52 of Year 5: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5 |  | 0.0 (NA) — SD was not estimable for 1 participant.
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change from Baseline in the NIS Component: Cranial Nerves Score Score at Week 52 of Year 4; Test type: Superiority; p = 0.941, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -0.01, 95% CI 2-sided [-0.19 to 0.17]

16. Secondary Outcome: Change From Baseline in the NIS Component: Muscle Weakness Score at Week 52 of Years 4 and 5
Description: Muscle weakness involves testing 19 movements of muscles. The score range of this component is 0 to 152 points. Higher scores indicate worsening. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Week 52 of Years 4 and 5
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 9 | 14
score on a scale
  Change From Baseline at Week 52 of Year 4 | 23.67 (16.712) | 14.71 (19.479)
  Change From Baseline at Week 52 of Year 5: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5 |  | 13.75 (NA) — SD was not estimable for 1 participant.
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change from Baseline in the NIS Component: Muscle Weakness Score at Week 52 of Years 4; Test type: Superiority; p = 0.011, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -9.56, 95% CI 2-sided [-16.97 to -2.16]

17. Secondary Outcome: Change From Baseline in the NIS Component: Reflexes Score at Week 52 of Years 4 and 5
Description: The Reflexes Score involves testing 5 reflexes to stimuli. The score range of this component is 0 to 20 points. Higher scores indicate worsening. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Week 52 of Years 4 and 5
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 9 | 14
score on a scale
  Change From Baseline at Week 52 of Year 4 | 4.17 (3.553) | 2.32 (1.957)
  Change From Baseline at Week 52 of Year 5: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5 |  | 4.00 (NA) — SD was not estimable for 1 participant.
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change from Baseline in the NIS Component: Reflexes Score at Week 52 of Years 4; Test type: Superiority; p = 0.356, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -1.05, 95% CI 2-sided [-3.28 to 1.18]

18. Secondary Outcome: Change From Baseline in the NIS Component: Sensory Score at Week 52 of Years 4 and 5
Description: The Sensory Score is based on testing an index finger and a big toe each to 4 stimuli. The score of this component ranges from 0 to 32 points. Higher scores indicate impairment. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Week 52 of Years 4 and 5
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 9 | 14
score on a scale
  Change From Baseline at Week 52 of Year 4 | 7.94 (5.288) | 1.29 (3.662)
  Change From Baseline at Week 52 of Year 5: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5 |  | 0.00 (NA) — SD was not estimable for 1 participant.
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change from Baseline in the NIS Component: Sensory Score at Week 52 of Years 4; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -5.38, 95% CI 2-sided [-8.58 to -2.19]

19. Secondary Outcome: Change From Baseline in the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) Questionnaire Total Score at Weeks 78 and 156
Description: The Norfolk QoL-DN score is a measure of physical function/large fiber neuropathy, symptoms, activities of daily living, small fiber neuropathy, and autonomic neuropathy. The Norfolk QoL-DN total score has a range of -4 to 136, and a higher Norfolk QoL-DN score indicates poorer QoL. A positive change from Baseline indicates worsening in the QoL. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156 and at the end of each subsequent treatment year (Week 52 of Years 4 and 5)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
score on a scale
  Change From Baseline at Week 78: number analyzed (Participants) | 34 | 71
  Change From Baseline at Week 78 | 15.22 (24.024) | 3.76 (20.832)
  Change From Baseline at Week 156: number analyzed (Participants) | 22 | 41
  Change From Baseline at Week 156 | 14.94 (28.944) | 5.98 (22.891)
  Change From Baseline at Week 52 of Year 4: number analyzed (Participants) | 9 | 14
  Change From Baseline at Week 52 of Year 4 | 6.22 (18.600) | 2.36 (25.120)
  Change From Baseline at Week 52 of Year 5: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5 |  | -1.00 (NA) — SD was not estimable for 1 participant.
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the Norfolk QOL-DN Questionnaire Total Score at Week 78; Test type: Superiority; p = 0.026, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -9.31, 95% CI 2-sided [-17.48 to -1.14]
Statistical Analysis 2: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the Norfolk QOL-DN Questionnaire Total Score at Week 156; Test type: Superiority; p = 0.107, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -7.40, 95% CI 2-sided [-16.41 to 1.62]
Statistical Analysis 3: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the Norfolk QOL-DN Questionnaire Total Score at Week 52 of Year 4; Test type: Superiority; p = 0.669, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -2.72, 95% CI 2-sided [-15.22 to 9.77]

20. Secondary Outcome: Change From Baseline in the Norfolk QoL-DN Physical Functioning/Large Fiber Neuropathy Domain Score
Description: The Norfolk QoL-DN physical functioning/large fiber neuropathy domain score is a sub-score of the total Norfolk QoL-DN Questionnaire. The Norfolk QoL-DN physical function/large fiber neuropathy domain score has a range of -4 to 56, and a higher Norfolk QoL-DN domain score indicates poorer quality of life (QoL). A positive change from Baseline indicates worsening in the QoL. MMRM was used for the analysis.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156 and at the Week 52 of Year 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 18 | 26
score on a scale
  Change From Baseline at Week 78: number analyzed (Participants) | 14 | 23
  Change From Baseline at Week 78 | 11.21 (11.026) | 3.61 (11.500)
  Change From Baseline at Week 156: number analyzed (Participants) | 5 | 11
  Change From Baseline at Week 156 | 12.60 (10.784) | -0.55 (8.042)
  Change From Baseline at Week 52 of Year 4: number analyzed (Participants) | 2 | 4
  Change From Baseline at Week 52 of Year 4 | 9.50 (9.192) | 3.50 (7.047)
Statistical Analysis 1: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the Norfolk QOL-DN Change From CS2 Baseline in the Norfolk QOL-DN Questionnaire Total Score at Week 78; Test type: Superiority; p = 0.097, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -6.30, 95% CI 2-sided [-13.75 to 1.15]
Statistical Analysis 2: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change from Baseline in the Norfolk QoL-DN Physical Functioning/Large Fiber Neuropathy Domain Score at Week 156; Test type: Superiority; p = 0.081, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -8.89, 95% CI 2-sided [-18.88 to 1.11]
Statistical Analysis 3: Comparison: Previous Placebo-Inotersen 300 mg vs Previous Inotersen-Inotersen 300 mg; Change From Baseline in the Norfolk QOL-DN Physical Functioning/Large Fiber Neuropathy Domain Score at Week 52 of Year 4; Test type: Superiority; p = 0.171, MMRM — [p-value comment as in outcome 9, analysis 1]; Least Squares Mean Difference = -11.87, 95% CI 2-sided [-28.89 to 5.16]

21. Secondary Outcome: Change From Baseline in the Modified Body Mass Index (mBMI) at Weeks 78 and 156
Description: BMI=weight (kg)/[height (m)^2]. The mBMI is the BMI multiplied by the serum albumin (g/L).
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kg/m^2*g/L
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
kg/m^2*g/L
  Change From Baseline at Week 78: number analyzed (Participants) | 35 | 71
  Change From Baseline at Week 78 | -166.27 (159.644) | -161.52 (134.779)
  Change From Baseline at Week 156: number analyzed (Participants) | 21 | 39
  Change From Baseline at Week 156 | -191.68 (130.370) | -172.52 (131.602)

22. Secondary Outcome: Change From Baseline in the Body Mass Index (BMI) at Weeks 78 and 156
Description: BMI=weight (kg)/[height (m)^2].
Time Frame: Baseline, Weeks 78 and 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
kg/m^2
  Change From Baseline at Week 78: number analyzed (Participants) | 35 | 71
  Change From Baseline at Week 78 | -0.16 (2.617) | -0.44 (1.427)
  Change From Baseline at Week 156: number analyzed (Participants) | 21 | 39
  Change From Baseline at Week 156 | -0.34 (1.908) | -0.66 (2.220)

23. Secondary Outcome: Percentage of Participants With Change From Baseline in the Polyneuropathy Disability (PND) Score
Description: PND score is defined as I = sensory disturbances in limbs without motor impairment; II = difficulty walking without the need of a walking aid; III = one stick or one crutch required for walking; IV = two sticks or two crutches needed. V = wheelchair required or patient confined to bed. The change from Baseline values have been categorized as: improved, not changed, worsened, and unknown. Percentage of participants with changes from Baseline are presented category-wise in this outcome measure. Only categories with at least one participant with event are reported.
Time Frame: Baseline, Weeks 78 and 156 and at the end of each subsequent treatment year (Week 52 of each year)
Population: FAS included all enrolled participants who received at least 1 injection of inotersen in this study (CS3) and who had at least 1 post-baseline efficacy assessment for the mNIS+7 score or Norfolk QoL-DN questionnaire total score collected after CS3 Study Day 1. Number analyzed is the number of participants with data available for analysis at the given time point for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
percentage of participants
  Change From Baseline at Week 78: Improved: number analyzed (Participants) | 36 | 71
  Change From Baseline at Week 78: Improved | 5.6 | 11.3
  Change From Baseline at Week 78: Not Changed: number analyzed (Participants) | 36 | 71
  Change From Baseline at Week 78: Not Changed | 69.4 | 62.0
  Change From Baseline at Week 78: Worsened: number analyzed (Participants) | 36 | 71
  Change From Baseline at Week 78: Worsened | 25.0 | 26.8
  Change From Baseline at Week 156: Improved: number analyzed (Participants) | 21 | 41
  Change From Baseline at Week 156: Improved | 4.8 | 7.3
  Change From Baseline at Week 156: Not Changed: number analyzed (Participants) | 21 | 41
  Change From Baseline at Week 156: Not Changed | 52.4 | 56.1
  Change From Baseline at Week 156: Worsened: number analyzed (Participants) | 21 | 41
  Change From Baseline at Week 156: Worsened | 42.9 | 36.6
  Change From Baseline at Week 52 of Year 4: Improved: number analyzed (Participants) | 9 | 14
  Change From Baseline at Week 52 of Year 4: Improved | 11.1 | 14.3
  Change From Baseline at Week 52 of Year 4: Not Changed: number analyzed (Participants) | 9 | 14
  Change From Baseline at Week 52 of Year 4: Not Changed | 33.3 | 42.9
  Change From Baseline at Week 52 of Year 4: Worsened: number analyzed (Participants) | 9 | 14
  Change From Baseline at Week 52 of Year 4: Worsened | 55.6 | 42.9
  Change From Baseline at Week 52 of Year 5: Not Changed: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5: Not Changed |  | 100

24. Secondary Outcome: Percent Change From Baseline in Global Longitudinal Strain (GLS) by Echocardiogram (ECHO) in the Cardiomyopathy-ECHO (CM-ECHO) Set
Description: GLS by ECHO is a measure of cardiac systolic function.
Time Frame: Baseline, Weeks 78 and 156
Population: The Cardiomyopathy-echocardiogram (CM-ECHO) Set included the subset of the 420915-CS2 Randomized Set that had a diagnosis of transthyretin (TTR) cardiomyopathy at study entry of the parent study, but were not in the ECHO Subgroup in the parent study, plus participants who qualified to participate in the ECHO Subgroup (whether consented or not). Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 27 | 52
percent change
  Change From Baseline at Week 78: number analyzed (Participants) | 18 | 32
  Change From Baseline at Week 78 | 0.38 (3.178) | -0.74 (3.120)
  Change From Baseline at Week 156: number analyzed (Participants) | 9 | 20
  Change From Baseline at Week 156 | 1.46 (5.313) | 0.07 (4.318)

25. Secondary Outcome: Percent Change From Baseline in GLS by ECHO in the CS3 ECHO Subgroup
Description: GLS by ECHO is a measure of cardiac systolic function.
Time Frame: Weeks 78 and 156
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 17 | 30
percent change
  Percent Change From Baseline at Week 78: number analyzed (Participants) | 12 | 18
  Percent Change From Baseline at Week 78 | -6.93 (20.232) | 8.99 (26.201)
  Percent Change From Baseline at Week 156: number analyzed (Participants) | 5 | 12
  Percent Change From Baseline at Week 156 | -2.79 (24.580) | 11.46 (29.383)

26. Secondary Outcome: Change From Baseline in Transthyretin (TTR) Level
Description: Transthyretin protein concentration in serum was measured.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
g/L
  Change From Baseline at Week 78: number analyzed (Participants) | 36 | 72
  Change From Baseline at Week 78 | -0.1581 (0.05887) | -0.1555 (0.06751)
  Change From Baseline at Week 156: number analyzed (Participants) | 25 | 43
  Change From Baseline at Week 156 | -0.1498 (0.06366) | -0.1692 (0.06025)

27. Secondary Outcome: Change From Baseline in Retinol Binding Protein 4 (RBP4) Level
Description: RBP4 protein concentration in serum was measured.
Time Frame: Baseline (Baseline is the Baseline of the Previous Study- Study CS2), Weeks 78 and 156, and at the end of each subsequent treatment year (Week 52 of Years 4 and 5)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: micrograms per liter (µg/L)
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 81
micrograms per liter (µg/L)
  Change From Baseline at Week 78: number analyzed (Participants) | 36 | 72
  Change From Baseline at Week 78 | -21073.1 (11038.53) | -19365.9 (10511.83)
  Change From Baseline at Week 156: number analyzed (Participants) | 25 | 43
  Change From Baseline at Week 156 | -21489.4 (10670.52) | -22372.3 (10372.05)
  Change From Baseline at Week 52 of Year 4: number analyzed (Participants) | 9 | 14
  Change From Baseline at Week 52 of Year 4 | -28307.1 (9539.75) | -24893.7 (5559.01)
  Change From Baseline at Week 52 of Year 5: number analyzed (Participants) | 0 | 1
  Change From Baseline at Week 52 of Year 5 |  | -24444.0 (NA) — SD was not estimable for 1 participant.

28. Secondary Outcome: Ctrough: Trough Plasma Concentration of ISIS 420915
Time Frame: Pre-dose on Days 1, 43, 85, 120, 176, 267, 358, 449, 540, 631, 722, 813, 904, 995, 1086, 1268; Days 1359 and 1450 of Year 4; Days 1632, 1723 and 1814 of Year 5
Population: CS3 Pharmacokinetic (PK) Set included all enrolled participants who received at least 1 dose of inotersen in CS3 and who had at least 1 evaluable PK sample collected and analyzed with reportable result in CS3. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
Number analyzed (Participants) | 50 | 85
nanograms per milliliter (ng/ml)
  Day 1: number analyzed (Participants) | 49 | 83
  Day 1 | NA (NA) — The data was below the lower limit of quantification (LLOQ), hence the geometric mean and geometric coefficient of variation were not estimable. | 34.1 (247)
  Day 43: number analyzed (Participants) | 41 | 63
  Day 43 | 22.9 (97.6) | 74.0 (123)
  Day 85: number analyzed (Participants) | 37 | 58
  Day 85 | 28.6 (43.6) | 83.0 (138)
  Day 120: number analyzed (Participants) | 27 | 31
  Day 120 | 31.5 (43.7) | 81.9 (142)
  Day 176: number analyzed (Participants) | 36 | 52
  Day 176 | 38.0 (52.9) | 80.0 (104)
  Day 267: number analyzed (Participants) | 24 | 41
  Day 267 | 47.3 (83.4) | 98.2 (183)
  Day 358: number analyzed (Participants) | 26 | 48
  Day 358 | 56.2 (102) | 110 (130)
  Day 449: number analyzed (Participants) | 25 | 37
  Day 449 | 71.1 (158) | 130 (218)
  Day 540: number analyzed (Participants) | 26 | 39
  Day 540 | 78.7 (163) | 111 (219)
  Day 631: number analyzed (Participants) | 19 | 28
  Day 631 | 83.8 (211) | 141 (187)
  Day 722: number analyzed (Participants) | 26 | 32
  Day 722 | 97.6 (245) | 101 (127)
  Day 813: number analyzed (Participants) | 14 | 28
  Day 813 | 98.0 (354) | 150 (273)
  Day 904: number analyzed (Participants) | 11 | 27
  Day 904 | 91.4 (230) | 116 (148)
  Day 995: number analyzed (Participants) | 12 | 15
  Day 995 | 147 (809) | 134 (246)
  Day 1086: number analyzed (Participants) | 13 | 27
  Day 1086 | 131 (340) | 101 (159)
  Day 1268 of Year 4: number analyzed (Participants) | 13 | 16
  Day 1268 of Year 4 | 167 (258) | 102 (202)
  Day 1359 of Year 4: number analyzed (Participants) | 4 | 10
  Day 1359 of Year 4 | 432 (307) | 157 (233)
  Day 1450 of Year 4: number analyzed (Participants) | 4 | 8
  Day 1450 of Year 4 | 55.0 (61.1) | 83.0 (111)
  Day 1632 of Year 5: number analyzed (Participants) | 1 | 4
  Day 1632 of Year 5 | 37.4 (NA) — The data was below the LLOQ, hence the geometric coefficient of variation was not estimable. | 75.3 (26.9)
  Day 1723 of Year 5: number analyzed (Participants) | 1 | 0
  Day 1723 of Year 5 | 113 (NA) — The data was below the LLOQ, hence the geometric coefficient of variation was not estimable. |
  Day 1814 of Year 5: number analyzed (Participants) | 0 | 1
  Day 1814 of Year 5 |  | 62.1 (NA) — The data was below the LLOQ, hence the geometric coefficient of variation was not estimable.

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 3 months post treatment period of 260 weeks (Up to approximately 272 weeks)
Description: SS included all enrolled participants who received at least 1 injection of inotersen in CS3.
Groups:
- Previous Placebo-Inotersen 300 mg: Participants received SC doses of 300 mg inotersen once weekly for up to 260 weeks. Participants who received inotersen-matching placebo in ISIS 420915-CS2 study were included in this group.
- Previous Inotersen-Inotersen 300 mg: Participants received SC doses of 300 mg inotersen once weekly for up to 260 weeks. Participants who received inotersen in ISIS 420915-CS2 study were included in this group.
Arm/Group | Previous Placebo-Inotersen 300 mg | Previous Inotersen-Inotersen 300 mg
All-Cause Mortality (participants affected / at risk) | 2/50 | 15/85
Serious Adverse Events (participants affected / at risk) | 18/50 | 46/85
Other Adverse Events (participants affected / at risk) | 50/50 | 80/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Placebo-Inotersen 300 mg (N=50) | Previous Inotersen-Inotersen 300 mg (N=85)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 4
Cardiac failure (Cardiac disorders) | 2 | 3
Cardiac failure acute (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Corneal perforation (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal hypomotility (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Cellulitis (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial toxaemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis streptococcal (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Measles (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spleen contusion (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 2
Calculus bladder (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Ovarian mass (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Previous Placebo-Inotersen 300 mg (N=50) | Previous Inotersen-Inotersen 300 mg (N=85)
Nausea (Gastrointestinal disorders) | 8 | 25
Diarrhoea (Gastrointestinal disorders) | 13 | 21
Fatigue (General disorders) | 7 | 20
Urinary tract infection (Infections and infestations) | 13 | 18
Fall (Injury, poisoning and procedural complications) | 11 | 18
Vomiting (Gastrointestinal disorders) | 8 | 16
Chills (General disorders) | 7 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 16
Oedema peripheral (General disorders) | 9 | 13
Injection site pain (General disorders) | 6 | 12
Pyrexia (General disorders) | 2 | 11
Injection site erythema (General disorders) | 4 | 12
Constipation (Gastrointestinal disorders) | 4 | 12
Syncope (Nervous system disorders) | 4 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 10
Abdominal pain (Gastrointestinal disorders) | 1 | 8
Anaemia (Blood and lymphatic system disorders) | 5 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Orthostatic hypotension (Vascular disorders) | 4 | 7
Hypotension (Vascular disorders) | 1 | 7
Headache (Nervous system disorders) | 7 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Dizziness (Nervous system disorders) | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7
Hypertension (Vascular disorders) | 1 | 5
Nasopharyngitis (Infections and infestations) | 3 | 7
Injection site pruritus (General disorders) | 3 | 7
Weight decreased (Investigations) | 4 | 7
Hypoaesthesia (Nervous system disorders) | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Asthenia (General disorders) | 4 | 6
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 | 6
Paraesthesia (Nervous system disorders) | 4 | 6
Insomnia (Psychiatric disorders) | 0 | 6
Haematuria (Renal and urinary disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
Bronchitis (Infections and infestations) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 5
Atrial fibrillation (Cardiac disorders) | 4 | 5
Balance disorder (Nervous system disorders) | 1 | 5
Injection site rash (General disorders) | 4 | 5
Oedema (General disorders) | 2 | 5
Platelet count decreased (Investigations) | 1 | 5
Sinusitis (Infections and infestations) | 2 | 5
Urinary retention (Renal and urinary disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Influenza (Infections and infestations) | 4 | 4
Cataract (Eye disorders) | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4
Gait disturbance (General disorders) | 3 | 4
Glomerular filtration rate decreased (Investigations) | 4 | 4
Injection site bruising (General disorders) | 4 | 4
Influenza like illness (General disorders) | 5 | 3
Dry eye (Eye disorders) | 3 | 3
Herpes zoster (Infections and infestations) | 4 | 3
Cellulitis (Infections and infestations) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Wound (Injury, poisoning and procedural complications) | 3 | 1
Pneumonia (Infections and infestations) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02175004/Prot_SAP_000.pdf